CLINICAL TRIAL: NCT02273843
Title: Effect of Different Dosages Oral Vitamin D on Serum Interleukin-6 in Preterm Infants With Late-onset Sepsis
Brief Title: A Trial on Different Dosages of Vitamin D in Preterm Infants With Late-onset Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Hesham Abdel-Hady, Professor of Pediatrics, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS 306
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Prematurity; Late-onset Sepsis
Keywords: Preterm; late-onset sepsis; Vitamin D; Dose; Interleukin-6; Tumor necrosis factor-alpha
MeSH Terms: conditions — Premature Birth | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-dose vitamin D (Experimental): Will receive oral cholecalciferol (vitamin D3) in a single daily dose of 800 IU from the time of diagnosis of sepsis until discharge from the NICU
  Interventions: Drug: High-dose vitamin D 3
- Conventional-dose vitamin D (Active Comparator): Will receive oral cholecalciferol (vitamin D3) in a single daily dose of 400 IU from the time of diagnosis of sepsis until discharge from the NICU
  Interventions: Drug: Conventional-Dose Vitamin D 3

INTERVENTIONS:
Drug: High-dose vitamin D 3 — Will receive oral cholecalciferol (vitamin D3) in a single daily dose of 800 IU from the time of diagnosis of sepsis until discharge from the NICU
  Other Names: High-dose cholecalciferol
  Arms: High-dose vitamin D
Drug: Conventional-Dose Vitamin D 3 — Will receive oral cholecalciferol (vitamin D3) in a single daily dose of 400 IU from the time of diagnosis of sepsis until discharge from the NICU
  Other Names: Conventional-dose cholecalciferol
  Arms: Conventional-dose vitamin D

SUMMARY:
This is a randomized controlled trial (RCT) to evaluate the influence of different doses of vitamin D3 (800 IU/d versus 400 IU/d), on serum levels of interleukin (IL)-6, TNF-alpha and C- reactive (CRP) in premature infants with clinical evidence of late-onset sepsis and to assess its influence on clinical outcomes of these infants.

DETAILED DESCRIPTION:
Vitamin D has an important role in the regulation of both the innate and adaptive immune systems. There are very few studies of such roles in the neonatal population. It is potentially an attractive therapeutic agent for sepsis given its low cost and low risk of toxicity and side effects. There is no consensus regarding to the dose of vitamin D supplementation required for preterm infants given the paucity of evidence. AAP and ESPGHAN have recommended different dosages of vitamin D ranging from 400 IU to 1000 IU per day. The influence of different doses of vitamin D on immunological status and clinical outcomes of preterm infants with late-onset sepsis has not been evaluated before. This RCT will evaluate the influence of different doses of vitamin D3 (800 IU/d versus 400 IU/d), on serum levels of interleukin (IL)-6, TNF-alpha and C- reactive (CRP) in premature infants with clinical evidence of late-onset sepsis we will also evaluate their safety and influence on clinical outcomes of these infants

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants (28-37 wk gestational age)
* Late-onset sepsis defined as clinical signs suggestive of infection after 72 h of birth. Clinical sepsis will be defined as the presence of three or more of the following categories of clinical signs:

  1. Temperature instability (hypothermia, hyperthermia);
  2. Respiratory (grunting, intercoastal retraction, apnea, tachypnea, cyanosis);
  3. Neurologic (hypotonia, lethargy, seizures);
  4. Gastrointestinal (feeding intolerance, abdominal distension).

Exclusion Criteria:

* Major congenital anomalies.
* Chromosomal anomalies.
* Known inborn error(s) of metabolism

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Serum interleukin-6 | At trial entry and 7 days after daily vitamin D supplementation therapy
  Serum levels of interleukin-6 (IL-6) will be evaluated at enrollment and 7 days after daily vitamin D supplementation therapy. IL-6 concentrations will be determined by Endogenous Interleukin-ELISA
Serum tumor necrosis-alpha | At trial entry and 7 days after daily vitamin D supplementation therapy
  Serum levels of tumor necrosis-alpha (TNF-alpha) will be evaluated at enrollment and 7 days after daily vitamin D supplementation therapy

SECONDARY OUTCOMES:
Serum C-reactive protein (CRP) | At trial entery and 7 days after daily vitamin D supplementation therapy
  Serum CRP will be evaluated at enrollment and 7 days
Serum 25(OH)D levels | at trial entry, 7 days after daily vitamin D supplementation therapy and at 40 weeks postmenstrual age
  Serum 25(OH)D levels will be measured by ELISA at trial entry, at day 7 and at 40 weeks postmenstrual age
Serum calcium, phosphorus and urinary calcium | Participants will be followed for the duration of hospital stay, serum calcium, phosphorus and urinary calcium well be assessed every week for an expected average of 5 weeks
  Participants will be followed for the duration of hospital stay, serum calcium, phosphorus and urinary calcium well be assessed every week for an expected average of 5 weeks
Abdominal ultrasonography | 40 weeks postmenstrual age
  Abdominal ultrasonography to detect any nephrocalcinosis will be done at 40 weeks postmenstrual age
Mortality | Baseline
  In-hospital mortality during NICU admission for an expected average of 5 weeks
Neonatal morbidities | Participants will be followed for the duration of hospital stay, for an expected average of 4 weeks
  Participants will be followed for the duration of hospital stay, for an expected average of 5 weeks and the incidence of neonatal morbidities e.g. NEC, retinopathy of prematurity, disseminated intravascular coagulopathy and renal dysfunction will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Unit, Mansoura University Children Hospital, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Moromizato T, Litonjua AA, Braun AB, Gibbons FK, Giovannucci E, Christopher KB. Association of low serum 25-hydroxyvitamin D levels and sepsis in the critically ill. Crit Care Med. 2014 Jan;42(1):97-107. doi: 10.1097/CCM.0b013e31829eb7af. PMID 23982028
- [Background] Hewison M. Vitamin D and the immune system: new perspectives on an old theme. Endocrinol Metab Clin North Am. 2010 Jun;39(2):365-79, table of contents. doi: 10.1016/j.ecl.2010.02.010. PMID 20511058
- [Background] Kim SY. The pleiomorphic actions of vitamin D and its importance for children. Ann Pediatr Endocrinol Metab. 2013 Jun;18(2):45-54. doi: 10.6065/apem.2013.18.2.45. Epub 2013 Jun 30. PMID 24904851
- [Background] Agostoni C, Buonocore G, Carnielli VP, De Curtis M, Darmaun D, Decsi T, Domellof M, Embleton ND, Fusch C, Genzel-Boroviczeny O, Goulet O, Kalhan SC, Kolacek S, Koletzko B, Lapillonne A, Mihatsch W, Moreno L, Neu J, Poindexter B, Puntis J, Putet G, Rigo J, Riskin A, Salle B, Sauer P, Shamir R, Szajewska H, Thureen P, Turck D, van Goudoever JB, Ziegler EE; ESPGHAN Committee on Nutrition. Enteral nutrient supply for preterm infants: commentary from the European Society of Paediatric Gastroenterology, Hepatology and Nutrition Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2010 Jan;50(1):85-91. doi: 10.1097/MPG.0b013e3181adaee0. PMID 19881390
- [Background] Abrams SA; Committee on Nutrition. Calcium and vitamin d requirements of enterally fed preterm infants. Pediatrics. 2013 May;131(5):e1676-83. doi: 10.1542/peds.2013-0420. Epub 2013 Apr 29. PMID 23629620
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Abdel-Hady H, Yahia S, Megahed A, Mosbah A, Seif B, Nageh E, Bhattacharjee I, Aly H. Mediators in Preterm Infants With Late-onset Sepsis: A Randomized Controlled Trial. J Pediatr Gastroenterol Nutr. 2019 Apr;68(4):578-584. doi: 10.1097/MPG.0000000000002238. PMID 30896608